CLINICAL TRIAL: NCT03010345
Title: The Use of Self Inflating Tissue Expanders In The Treatment Of Alveolar Cleft
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Hany shams, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo university kasr el ainy
Record Dates: First submitted 2016-12-27; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Cleft of Alveolar Ridge

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osmed self inflating tissue expanders (Experimental): All patients will undergo a two-stage procedure ,second stage under General endotracheal anesthesia. The first stage will be placement of the expanders. The second stage will be 21 days later, with removal of the expanders, palatal revision, and closure of the oronasal fistula
  Interventions: Device: Osmed self inflating tissue expanders
- Iliac bone graft (Experimental): Placement of bone graft without the use of self inflating expanders
  Interventions: Other: Iliac bone graft

INTERVENTIONS:
Device: Osmed self inflating tissue expanders — Osmed self inflating tissue expanders will be placed 21 days before bone grafting the cleft to gain soft tissue coverage
  Arms: Osmed self inflating tissue expanders
Other: Iliac bone graft — Bone grafting the cleft without the use of osmed self inflating tissue expander
  Arms: Iliac bone graft

SUMMARY:
patient receiving treatment using the osmed expander will have enough soft tissue coverage securing the bone graft which will be placed in a later stage to close the alveolar cleft.

DETAILED DESCRIPTION:
to prove that the group treated with osmed expanders will suffer no soft tissue dehiscence and will have a higher volume of soft tissue at the stage of bone grafting.

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Patients suffering from alveolar cleft with anterior fistulas.
* Age Between 7 and 13 Years
* Both sexes.
* Patients physically able to tolerate surgical and restorative procedures. Good oral hygiene.
* Highly motivated patients.

Exclusion Criteria:

* non motivated patients

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome : Absence of nasal regurgitation. Binary (Yes/No) | 21 days

SECONDARY OUTCOMES:
Secondary Outcome : absence of soft tissue Dehiscence and preservation of bone graft volume , volume per cubic meter(Measured by cbct) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Galal El Behiry, Phd, Study Director — Cairo University
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No